CLINICAL TRIAL: NCT00313079
Title: A Phase I Study of mAb 216 With Chemotherapy for the Treatment of Adult Patients With Relapsed or Refractory B-Lineage Acute Lymphoblastic Leukemia
Brief Title: Monoclonal Antibody (mAb) 216 With Chemotherapy in Adult Relapsed or Refractory B-Lineage Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Steven E. Coutre (Other)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMALL0003; 96613 (Other: Stanford University alternate IRB Number)
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia, Lymphocytic; Leukemia; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MAb 216 — Dosage: 1.25mg/kg intravenous with dose escalation
  Other Names: Monoclonal Antibody 216
Drug: Vincristine — Dosage: 1.5mg/m2 intravenous weekly X 4
  Other Names: Oncovin; leurocristine; VCR

SUMMARY:
A phase I trial in patients with relapsed or refractory leukemia of a human monoclonal antibody that kills B cell acute lymphoblastic leukemia. Trial will study safety, pharmacokinetics, and anti tumor activity of the antibody given as a single agent and with vincristine.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Age Patients must be >= 18 years old at the time of study entry.

3.1.2 Diagnosis

3.1.2.1 Histologic Verification Patients must have had histologic verification of B-lineage ALL with bone marrow relapse or refractory disease that is unresponsive to traditional chemotherapy.

3.1.2.2 For patients WITHOUT prior allogeneic BMT:

1. Second or subsequent bone marrow relapse
2. Primary refractory marrow disease
3. M3 marrow (>25% blasts) or >25% leukemic blasts in peripheral blood

3.1.2.3 For patients WITH prior allogeneic BMT:

1. First or subsequent bone marrow relapse post-BMT
2. M3 marrow or M2 (>5 % and <25% blasts) if cytogenetic or VNTR confirmation

3.1.3 Confirmation of antibody reactivity 3.1.3.1 Patient's leukemic blasts (peripheral blood or marrow) must be documented to bind mAb 216 in vitro (Teng lab) 3.1.3.2 Patient's RBC documented to NOT express fetal "i" antigen and RBC shown to NOT bind mAb 216 in vitro (Teng lab)

3.1.4 Patient Must Not Be Eligible For Therapies of Higher Priority

3.1.5 Performance Level (See Appendix I) Karnofsky >= 50%

3.1.6 Life Expectancy Must be at least 8 weeks.

3.1.7 Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

1. Myelosuppressive chemotherapy: Must not have received within one week of entry onto this study.
2. Biologic, including monoclonal antibodies: At least 2 weeks since the completion of therapy with a biologic agent including monoclonal antibodies.
3. Hydroxyurea can be used up to 72 hours before study entry

3.1.8 Organ Function Requirements

3.1.8.1 Bone Marrow Function: 3.1.8.1.1 No hematologic criteria for WBC, Hgb or platelets 3.1.8.1.2 Patients with thrombocytopenia should be responsive to platelet transfusions and must not have uncontrolled bleeding.

3.1.8.2 Adequate Renal Function Defined As:

- A serum creatinine that is less than or equal to 2 x normal for age

3.1.8.3 Adequate Liver Function Defined As:

* Total bilirubin <= 2 x upper limit of normal (ULN) for age, and
* SGPT (ALT) <= 5 x upper limit of normal (ULN) for age

3.1.8.4 Adequate Cardiac Function Defined As:

* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by gated radionuclide study.

3.1.9 Regulatory

3.1.9.1 All patients must sign a written informed consent. 3.1.9.2 All institutional (IRB) and FDA requirements for human studies must be met.

Exclusion Criteria:

3.2.1 CNS 3 or refractory CNS leukemia

3.2.2 Isolated extramedullary relapse

3.2.3 Uncontrolled infection

3.2.4 Lack of mAb 216 binding to patient's leukemic blasts in vitro

3.2.5 Binding of mAb 216 to the "i" antigen on patient's erythrocytes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
In this phase I study the endpoint is the determination of the maximum tolerable dose without toxicity.

SECONDARY OUTCOMES:
A decrease in leukemic blasts. The study will be terminated if unacceptable doseSecondary endpoints are a decrease in leukemic blasts. The study will be terminated if unacceptable dose limiting toxicity is found. This is a phase I trial to study safety.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson N Teng, Sub-Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Liedtke M, Twist CJ, Medeiros BC, Gotlib JR, Berube C, Bieber MM, Bhat NM, Teng NN, Coutre SE. Phase I trial of a novel human monoclonal antibody mAb216 in patients with relapsed or refractory B-cell acute lymphoblastic leukemia. Haematologica. 2012 Jan;97(1):30-7. doi: 10.3324/haematol.2011.045997. Epub 2011 Oct 11. PMID 21993685